CLINICAL TRIAL: NCT03730545
Title: Effect of Enteral Immunonutrition on Immune, Inflammatory Markers and Nutritional Status in Patients Undergoing Gastrectomy for Gastric Cancer：a Randomized Double Blinded Controlled Trial
Brief Title: Effect of Enteral Immunonutrition on Immune, Inflammatory Markers and Nutritional Status in Patients Undergoing Gastrectomy for Gastric Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yong Zhou, associate chief physician, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 396312366
Record Dates: First submitted 2018-10-25; First posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Gastric Cancer; Enteral Immunonutrition
Keywords: gastric cancer; enteral nutrition; enteral immunonutrition; immune function; inflammation response
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients were randomized to receive enteral immunonutrition or standard enteral nutrition in postoperative day 1 by enteral feeding.
Who Masked: Participant, Investigator
Masking Description: Eligible patients were randomly assigned in equal numbers to undergo SEN or EIN according to a computer-generated randomization list managed by a dietary nurse not involved in the study. The study was double-blind: SEN and EIN feeds were identical in color and type of container, so treatment assignments were not revealed to patients or to any staff members.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EIN group (Experimental): Enteral formula including not only basic energy components, but also immune components such as omega-3 fatty acids, glutamine (Gln), arginine (Arg), and nucleotide.
  Interventions: Dietary Supplement: enteral immunonutrition
- SEN group (Active Comparator): Enteral formula including only basic energy components.
  Interventions: Dietary Supplement: enteral immunonutrition

INTERVENTIONS:
Dietary Supplement: enteral immunonutrition — Enteral nutrition was started within 12h at an infusion rate of 20ml per hour for SEN group and 16ml per hour for EIN group in the first 24h. The rates of flow were gradually increasing with 50ml/h in SEN versus 40ml/h in EIN on day 2, 70ml/h versus 56ml/h on day 3 and 100ml/h versus 80ml/h until the 7th day depending on the feeding tolerance.

SUMMARY:
Enteral immunonutrition (EIN) has been gaining increasing attention, but data of its immune and anti-inflammatory function in patients undergoing gastrectomy for gastric cancer are poorly investigated. The aim of this study was to assess the effect of EIN on immune function, inflammation response and nutrition status when compared to standard enteral nutrition (SEN).

The investigators believe that the proportion of cluster of differentiation 4 T-cells(CD4＋T-cells), cluster of differentiation 3 T-cells(CD3＋T-cells) and the counts of CD4＋ / cluster of differentiation 8 T-cells (CD8＋), immunoglobulin G(IgG), immunoglobulin M(IgM), and immunoglobulin A (IgA) were larger in EIN group, while the level of WBC, CRP and TNF-α were lower and nutritional status was similar.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 80 years
* with histologically diagnosed cancer of stomach
* candidates for elective subtotal or total gastrectomy

Exclusion Criteria:

* pregnant or lactating woman,
* diagnoses of mental diseases
* resent severe concomitant diseases (chronic cardiopulmonary disease, chronic renal failure, etc.)
* known allergies to nutrition formula or component
* drug intolerance
* known immunodeficiency or autoimmune diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline serum level of immune cytokines to postoperative day 5 | baseline and postoperative day 5
  levels of IgA, IgG and IgM in g/L,
Change from baseline serum level of immune markers to postoperative day 5 | baseline, postoperative day 5(POD 5)
  count of CD4＋/CD8＋
Change from baseline serum concentration of immune markers to postoperative day 5 | baseline, postoperative day 5(POD 5)
  percentage of CD3＋ T cell of serum

SECONDARY OUTCOMES:
changes among baseline, postoperative day 1, 3 and 5 serum concentration of inflammatory markers | baseline, postoperative day 1, 3, and 5
  concentration of white blood cell (WBC), C-reactive protein (CRP), interleukin-6 (IL-6) in g/L, and levels of tumor necrosis factor-α (TNF-α) in ng/L
Change among baseline, postoperative day 3 and 5 serum nutritional markers | baseline,postoperative day 3 and 5
  concentration of albumin, prealbumin, and transferrin in g/L